CLINICAL TRIAL: NCT05925205
Title: Muscle Energy Technique Versus Strain Counterstrain in Treatment of Upper Trapezius Myofascial Pain Syndrome: A Double-Blinded Randomized Controlled Trial
Brief Title: Muscle Energy Technique Versus Strain Counterstrain for Upper Trapezius Myofascial Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Ibrahim, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T. 2023-2025
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Physical Therapy
Keywords: Muscle energy technique, strain counterstrain, trapezius.

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Firstly, the research assistant, another qualified physical therapist, performing the assessment process, pre and post-treatment, will be blinded regarding the patients allocation into the three treatment groups. Secondly, the patients themselves will be blinded regarding which treatment group they will be allocated into. So the research assistant won't know the randomization results, and the main investigator won't know the assessment results which will make it a double-blinded study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Experimental group 1.
  Interventions: Procedure: Muscle energy technique combined with the physical therapy program.
- Group B (Experimental): Experimental group 2.
  Interventions: Procedure: Strain counterstrain technique combined with the physical therapy program
- Group C (Experimental): Experimental group 3.
  Interventions: Procedure: The physical therapy program

INTERVENTIONS:
Procedure: Muscle energy technique combined with the physical therapy program. — A manual therapy technique
  Arms: Group A
Procedure: Strain counterstrain technique combined with the physical therapy program — A manual therapy technique
  Arms: Group B
Procedure: The physical therapy program — Electrotherapy and exercise.
  Arms: Group C

SUMMARY:
This study will be conducted to examine the superiority of effectiveness between muscle energy technique combined with physical therapy, strain counterstrain combined with physical therapy, and physical therapy alone in terms of pain intensity, pain pressure threshold, cervical lateral flexion and rotation range of motion, and neck function for patients with upper trapezius myofascial trigger points.

DETAILED DESCRIPTION:
Myofascial pain syndrome represents a common, overlooked, and under-diagnosed disorder that have very critical negative effects on people's lives. In addition, it overloads the societies and causes several burdens on healthcare systems. However, this disorder is usually dismissed by many clinicians keeping the patients in pain for long periods. The central feature of myofascial pain syndrome is the myofascial trigger points that when managed properly, the painful symptoms disappear. Muscle energy technique and strain counterstrain immediate effects were compared in a recent comparative study for patients with upper trapezius myofascial trigger points in terms of pain intensity, pain pressure threshold, and neck mobility. The results showed that there were improvements of both techniques with no significant differences between them. Regarding the evidence of the two techniques; muscle energy technique and strain counterstrain in the management of patients with upper trapezius myofascial trigger points, there is lack of high-quality evidence investigating the effectiveness and safety of both techniques for this population and there is a need for well-developed randomized controlled trial to take a step in the pyramid of levels of evidence for the use and applicability of them. After reviewing the available literature, it was found that there is no study directly combined both techniques with physical therapy protocol in a randomized clinical trial for patients with upper trapezius myofascial trigger points; this will enable us to compare the effects of them in a controlled design to examine and find out the differences between the three treatment protocols.

ELIGIBILITY:
Inclusion Criteria

Patients will be included in the study if they fulfil the following criteria:

1. They have active myofascial trigger points in the upper trapezius muscle bilaterally according to the established criteria for myofascial trigger points examination.
2. They have neck pain less than three months.
3. Their age ranges from 18 to 40 years old. Exclusion Criteria

Patients will be excluded from the study if they fulfil the following criteria:

1. Patients with chronic pain syndrome.
2. Patients having myofascial trigger points in other neck muscles.
3. Patients having a history of an injury or surgery or instability or deformity including both; cervical spine and shoulder.
4. Patients diagnosed with a neurological disorder including altered sensation, migraine, cervical spondylosis, radiculopathy, or myelopathy, and tumour.
5. Patients with a systemic disease including rheumatoid arthritis, Reiter's syndrome, diabetes, fibromyalgia syndrome, and severe medical or psychiatric disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-05-07 (Actual); Primary Completion 2024-05-07 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity. | Change from Baseline pain intensity at one month.
  Measurement of pain intensity using the visual analogue scale.
Change in the right side pain pressure threshold. | Change from Baseline right side pain pressure threshold at one month.
  Measurement of right side pain pressure threshold using the pressure algometer.
Change in the left side pain pressure threshold. | Change from Baseline left side pain pressure threshold at one month.
  Measurement of left side pain pressure threshold using the pressure algometer.
Change in cervical flexion range of motion. | Change from Baseline cervical flexion range of motion at one month.
  Measurement of cervical flexion range of motion using the cervical range of motion device.
Change in cervical extension range of motion. | Change from Baseline cervical extension range of motion at one month.
  Measurement of cervical extension range of motion using the cervical range of motion device.
Change in cervical right lateral flexion range of motion. | Change from Baseline cervical right lateral flexion range of motion at one month.
  Measurement of cervical right lateral flexion range of motion using the cervical range of motion device.
Change in cervical left lateral flexion range of motion. | Change from Baseline cervical left lateral flexion range of motion at one month.
  Measurement of cervical left lateral flexion range of motion using the cervical range of motion device.
Change in cervical right rotation range of motion. | Change from Baseline cervical right rotation range of motion at one month.
  Measurement of cervical right rotation range of motion using the cervical range of motion device.
Change in cervical left rotation range of motion. | Change from Baseline cervical left rotation range of motion at one month.
  Measurement of cervical left rotation range of motion using the cervical range of motion device.
Change in neck function. | Change from Baseline neck function at one month.
  Measurement of neck function using the neck disability index-Arabic version.

CONTACTS AND LOCATIONS:
Overall Officials: Bassem El Nahass, PhD, Study Director — Professor of Orthopaedic Physical Therapy, Faculty of Physical Therapy, Cairo University
Locations (1):
- The Outpatient Clinics, Faculty of Physical Therapy Kafrelsheikh University, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No